CLINICAL TRIAL: NCT00820976
Title: A Phase III, Randomized Multicenter Study of Induction With or Without Granulocyte Colony-Stimulating Factor in AML
Brief Title: Induction With or Without Granulocyte Colony-Stimulating Factor in AML Transplantation in AML
Acronym: TLG-AML-95-002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Turkish Leukemia Study Group (Other)
Responsible Party: Meral Beksac MD, principal investigator, Turkish Leukemia Sutdy Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLG-AML-95-002
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: AML
Keywords: G-CSF; AML; survival
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): remission induction with cytosine arabinoside amd idarubicine
- G-CSF (Experimental): G-CSF was administered starting on Day 8 until neutrophil recovery
  Interventions: Drug: G-CSF

INTERVENTIONS:
Drug: G-CSF — Filgrastim(5 µg/kg intravenously over 30 minutes ) was administered starting from day 8 until neutrophil recovery
  Other Names: Neupogen
  Arms: G-CSF

SUMMARY:
Background The effects of granulocyte colony-stimulating factors (G-CSF) on recovery following induction chemotherapy are widely accepted. However, their impact on response and survival has not been clarified yet. Male gender has been claimed to be a susceptibility factor for development of leukemia and shorten survival but effect of sex has not been analyzed in clinical trials utilizing G-CSF.

Design and Methods Efficacy and safety of G-CSF as an adjunct to de novo AML remission induction therapy was assessed in this prospective randomized Phase III multicenter trial. Patients were randomized to receive induction therapy consisting of either cytosine arabinoside 100mg/m2/d, days 1-10 and idarubicin 12 mg/m2/d, days 1-3 (control arm) or plus G-CSF (Filgrastim, 5 µg/kg/d starting from day 8 until absolute neutrophil count (ANC) over 0.5x109/L for two consecutive days) for a median duration of 14 days (G-CSF arm).

After achievement of CR, all patients received first consolidation course of Ara-C 1 gr/sq.m/d (d1-5) and Ida 12 mg/sq.m/d (d1-3). If patients did not have an HLA identical donor they were randomized to receive second course of consolidation either high dose Ara-C 3 gr/sq.m/d (d1, 3, 5) or G-CSF for collection of stem cells for the consecutive PBSCT.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML
* Age over 16
* Performance status greater than 60
* Previously untreated
* Peripheral blood white blood cell (WBC) count of less than (<) 0.5 x109/L, and/or marrow leukemic blasts< 20 % at 7th day of remission induction treatment

Exclusion Criteria:

* Previously treated
* Acute promyelocytic leukemia
* Age equal or younger than 15

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1996-03; Primary Completion 2000-03 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
response to induction | 3 year
overall survival | 3 year

REFERENCES:
- [Derived] Beksac M, Ali R, Ozcelik T, Ozcan M, Ozcebe O, Bayik M, Paydas S, Buyukasik Y, Ilhan O, Ozkalemkas F, Gurman G, Uysal A, Akan H, Soydan EA, Tunali A. Short and long term effects of granulocyte colony-stimulating factor during induction therapy in acute myeloid leukemia patients younger than 65: results of a randomized multicenter phase III trial. Leuk Res. 2011 Mar;35(3):340-5. doi: 10.1016/j.leukres.2010.07.005. Epub 2010 Jul 29. PMID 20673585